CLINICAL TRIAL: NCT03197883
Title: A Randomized, Evaluator-blind, Single-center and Two-arm Clinical Study Designed to Evaluate the Local Tolerance and Cosmetic Efficacy of a Topical Skin Care Formulation in Healthy Female Subjects With Mild to Advanced Photo-damaged Facial Skin Who Have Undergone a 70% Glycolic Acid Facial Peel Procedure
Brief Title: Assessment of the Cosmetic Benefit of a Skin Cream in Healthy Females With Mild to Advanced Photo-damaged Facial Skin Who Have Undergone a Glycolic Acid Facial Peel Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 206827
Record Dates: First submitted 2017-06-08; First posted 2017-06-23 (Actual); Results first posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-05

CONDITIONS: Skin Care
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants will apply a pea-sized quantity of test product (approximately 0.6-1 grams (g)) topically onto the fingertips and will apply twice daily (morning and evening) to the full face after cleansing. All participants will be instructed to continue using the facial cleanser twice-daily during the morning and evening and to apply the sunscreen in the morning (after application of test product) and at lunchtime.
  Interventions: Other: Test Product; Other: Cleanser; Other: Sunscreen
- Group 2 (Other): Participants will wet face with water and work a small amount of facial cleanser (approximately 0.6-1 g) into lather. Massage topically onto wet skin and rinse with water twice daily (morning and evening). After cleansing, participants will apply a pea-sized quantity (approximately 0.6-1 g) of the sunscreen in the morning and at lunchtime.
  Interventions: Other: Cleanser; Other: Sunscreen

INTERVENTIONS:
Other: Test Product — Restoring lipid balm
  Arms: Group 1
Other: Cleanser — Moisturizing facial cleanser
Other: Sunscreen — SPF (Sun Protection Factor) 50 sunscreen

SUMMARY:
To evaluate the local tolerance and cosmetic efficacy of a topical skin care formulation in healthy female participants with mild to advanced photo-damaged facial skin who have undergone a 70% Glycolic Acid facial peel procedure.

DETAILED DESCRIPTION:
This will be a randomized, evaluator-blind, single-center and two-arm clinical study designed to evaluate the local tolerance and cosmetic efficacy of a topical skin care formulation in healthy female participants with mild to advanced photo-damaged facial skin who have undergone a 70% Glycolic Acid facial peel procedure.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Females aged between 30 and 60 years inclusive.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical examination.
* Willingness to actively participate in the study and to attend all scheduled visits.
* Skin Type: Fitzpatrick phototype II-IV and participants with Glogau photoaging type II-III
* Females of childbearing potential who are, in the opinion of the investigator, practising a reliable method of contraception. Adequate contraception is defined as abstinence, oral contraceptive, either combined or progestogen alone or injectable progestogen or implants of levonorgestrel or estrogenic vaginal ring or percutaneous contraceptive patches or intrauterine device or intrauterine system or double barrier method (condom or occlusive cap [diaphragm or cervical vault caps] plus spermicidal agent [foam, gel, film, cream, suppository]) or male partner sterilization prior to the female participant's entry into the study, and this male is the sole partner for that participant.

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding.
* a) Active skin disease or open wound in the test area, b) Medical history of using a medicated acne treatment (e.g. Benzoyl Peroxide, Clindamycin, isotretinoin) within the last 24 months, c)Medical history of dysplastic nevi or melanoma, d) Preexisting inflammatory dermatoses such as psoriasis, atopic dermatitis, e) Moles, tattoos, scars, irritated skin, hairs, etc. at the test area that could, in the opinion of the investigator, influence the investigation, f) Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines within 7 days prior to screening and/or throughout the entire course of the study, g) Systemic use of over-the-counter (OTC) analgesics or anti-inflammatory drugs 24 hours prior to screening. h)Systemic use of any photosensitizing medication 2 weeks prior to screening, i) Intense sun exposure, UV-treatments or tanning salon visit within two weeks prior to screening, j) One of the following illnesses that might require regular systemic medication; Insulin-dependent diabetes, cancer, k) One of the following illnesses if not medicated: Asthma, hypertension, l) Medical history of abnormal response to sunlight, m) Participant's with a history of mental illness, n) Ocular surgery within the last 12 months.

  o) Ocular trauma, infection or inflammation within the last 3 months, p) Active blepharitis, conjunctivitis, uveitis, q) Any ocular pathology requiring topical ocular treatment within the last 1 month, r) Ocular laser within the last 3 months, s) Aesthetic, cosmetic or dermatological treatment in the treatment area (face), including the use of skin tone lightning products, within the last 3 months, t) Use of facial scrubs, depilatory creams, waxing and/or bleaching within the last 2 weeks prior to screening, u) Microdermabrasion and/or laser hair removal within the last 4 weeks prior to screening, v) Medical history of Herpes Simplex (Cold Sores).
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients and documented allergies to cosmetic products or study ingredients.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit and previous participation in this study.
* Recent history (within the last 5 years) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family.
* Required to work outside during daylight hours over the duration of the study and required or otherwise intending to spend prolonged periods of time outside during daylight hours over the duration of the study (e.g. holiday, sunbathing, and gardening).
* A score of "Severe" for any Dermatologist or Participant's Self-Assessed endpoint at any time for the study material sensitivity test.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Campinas, São Paulo, Brazil

REFERENCES:
- See also: Review and Approval was conducted on previous disclosure system and therefore, the document was uploaded directly to the PRS system. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=206827&attachmentIdentifier=86df9897-f813-4d6c-9249-1cd57a0baaec&fileName=gsk-206827-protocol-redact.pdf&versionIdentifier=
- See also: Review and Approval was conducted on previous disclosure system and therefore, the document was uploaded directly to the PRS system. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=206827&attachmentIdentifier=290500e9-fd13-4db3-a155-c5c1ef61ba57&fileName=gsk-206827-reporting-and-analysis-plan-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were recruited from one center in Brazil.
Pre-assignment Details: A total of 163 participants were screened, out of which 31 did not meet study criteria, 7 had adverse events (AEs), 1 participant was lost to follow-up, 1 withdrew his consent and 23 participants were not randomized in the study due to other reasons (not specified).
Groups:
- Test Product: Participants applied a pea-sized quantity of test product (approximately 0.6-1 grams (g)) topically onto the fingertips twice daily (morning and evening) to the full face after cleansing. All participants were instructed to continue using the facial cleanser twice-daily during the morning and evening and to apply the sunscreen in the morning (after application of test product) and at lunchtime.
- No Treatment: Participants had their face wet with water and a small amount of facial cleanser (approximately 0.6-1 g) into lather. It was massaged topically onto wet skin and rinsed with water twice daily (morning and evening). After cleansing, participants applied a pea-sized quantity (approximately 0.6-1 g) of the sunscreen in the morning and at lunchtime.
Period: Overall Study
Arm/Group | Test Product | No Treatment
Started | 50 | 50
Completed | 47 | 44
Not Completed | 3 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Other (Not Specified) | 0 | 5

BASELINE CHARACTERISTICS:
Population: The demographic characteristics has been reported for safety population (N=96). The safety population included all participants with at least 1 application of product in the test phase. This population was based on the treatment the participant actually received.
Groups:
- Test Product: Participants dispensed a pea-sized quantity of test product (approximately 0.6-1 g) onto the fingertips and applied twice daily (morning and evening) to the full face after cleansing. All participants were instructed to continue using the facial cleanser twice-daily during the morning and evening and to apply the sunscreen; approximately 0.6 to 1.0 g) on the full face in the morning (after application of test product) and at lunchtime.
- No Treatment: Participants dispensed approximately 0.6 to 1.0 g of cleanser into the hands, worked into a lather, massaged onto the full face (wet skin), and rinsed with water, twice a day (morning and evening). After cleansing, participants applied a pea-sized quantity (approximately 0.6-1 g) of the sunscreen in the morning and at lunchtime.
- Total: Total of all reporting groups
Arm/Group | Test Product | No Treatment | Total
Number analyzed (Participants) | 50 | 46 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (7.54) | 45.1 (8.35) | 45.5 (7.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 46 | 96
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 45 | 36 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I- Always Burns, Never Tans | 0 | 0 | 0
  II- Usually Burns, Tans Minimally | 16 | 15 | 31
  III- Sometimes mild Burn, Tans uniformly | 34 | 31 | 65
  IV- Burns Minimally, Always Tans well | 0 | 0 | 0
  V- Very rarely Burns, Tans very easily | 0 | 0 | 0
  VI- Never Burns, Never Tans | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Product Tolerability Based on Evaluator Global Assessment Scores
Description: The dermatologist assessed the local tolerance of the post-procedure skin care regimen in context of the expected effects of the procedure for each participant using the scale as below: 0 - Product regimen was well tolerated, 1 - product regimen was not well tolerated. The dermatologist observed on the total set of clinical and participant self-assessment data for each participant. Lower scale value implies that no clinically significant worsening of the expected signs/symptoms of the procedure, no new signs/symptoms manifest during product use. Whereas, higher scale value implies clear, clinically relevant worsening of the severity or frequency of expected signs/symptoms of the procedure and/or any occurrence of new, unexpected signs/symptoms during product use.
Time Frame: 14 days after completion of the facial peel procedure
Population: The safety population (N=96) included all participants with at least 1 application of product in test phase. This population was based on treatment the participant actually received. Of which, there were 50 in test product and 46 in no treatment. Number of participants (n=91) analyzed in this outcome measure signifies those who were evaluated.
Measure: Count of Participants; unit: Participants
Groups:
- Test Product: Participants applied a pea-sized quantity of test product (approximately 0.6-1 g) topically onto the fingertips twice daily (morning and evening) to the full face after cleansing. All participants were instructed to continue using the facial cleanser twice-daily during the morning and evening and to apply the sunscreen in the morning (after application of test product) and at lunchtime.
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 47 | 44
Participants
  Product was well tolerated | 47 | 44
  Product was not well tolerated | 0 | 0

2. Secondary Outcome: Change From Baseline in Total Score of Dermatologist Assessments
Description: The assessments of Erythema, Dryness, Desquamation and Edema were conducted by a dermatologist on the participant's skin condition at the 5 x 5 cm square area on the volar surface of forearm. The signs were scored on a scale. Erythema on 0-3 where, 0=none-no redness, 1=mild-slight redness, 2=moderate-definite redness, 3=severe-marked redness. Dryness on 0-3 where, 0=none-no dryness, 1=mild-barely perceptible, fine scales to limited areas of test site, 2=moderate-fine scales generalized to all areas of test site, 3=severe-scaling and peeling of skin over all areas of test site. Desquamation on 0-3 where, 0=none-no sign of peeling, 1=mild-barely perceptible scaling, 2=moderate-minimal scaling, 3=severe-moderate scaling. Edema on 0-3 where, 0=none-no edema, 1=mild-barely perceptible edema, 2=moderate-definite edema, 3=severe-pronounced edema. The measure is sum of participant scores, so a total score scale ranges from 0-12, with higher scores indicating increased signs of irritation.
Time Frame: 14 days after completion of the facial peel procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 50 | 46
Score on Scale
  At Baseline | 1.14 (0.904) | 1.00 (0.730)
  14 days after completion: number analyzed (Participants) | 47 | 44
  14 days after completion | 0.06 (0.438) | 0.09 (0.362)
  Change from Baseline at 14 days after completion: number analyzed (Participants) | 47 | 44
  Change from Baseline at 14 days after completion | -1.11 (0.814) | -0.86 (0.824)

3. Secondary Outcome: Number of Participants Reporting no/Mild/Moderate/Severe Change From Baseline in Individual Dermatologist Scores for Erythema, Edema, Desquamation and Dryness
Description: The signs/symptoms of participants were scored on a scale of 0 to 3 as below: Erythema: Score from 0=None-No evidence of erythema present, 1=Mild-Slight red coloration, 2=Moderate-Definite redness, 3=Severe-Marked erythema, bright red to dusky dark red in color. Dryness: Score from 0=None-No dryness, 1=Mild-Barely perceptible, fine scales or flakes present to limited areas of the test site, 2=Moderate-Fine scales or flakes generalized to all areas of the test site, 3=Severe -Scaling and peeling of skin over all areas of the test site. Desquamation score from 0=None-No evidence of desquamation/peeling, 1=Mild-Barely perceptible scaling; evident only on scratching, 2=Moderate-Minimal scaling, adherent to the skin, 3=Severe -Moderate scaling, loosely adherent to the skin and easily removable. Edema score from 0=None-No edema present, 1=Mild-Barely perceptible edema present, 2=Moderate-Definite edema present, 3=Severe-Marked/pronounced edema present.
Time Frame: 14 days after completion of the facial peel procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 47 | 44
Participants
  Erythema at 14 days after completion: None | 46 | 44
  Erythema at 14 days after completion: Mild | 1 | 0
  Erythema at 14 days after completion: Moderate | 0 | 0
  Erythema at 14 days after completion: Severe | 0 | 0
  Dryness at 14 days after completion: None | 46 | 41
  Dryness at 14 days after completion: Mild | 1 | 3
  Dryness at 14 days after completion: Moderate | 0 | 0
  Dryness at 14 days after completion: Severe | 0 | 0
  Desquamation at 14 days after completion: None | 46 | 43
  Desquamation at 14 days after completion: Mild | 1 | 1
  Desquamation at 14 days after completion: Moderate | 0 | 0
  Desquamation at 14 days after completion: Severe | 0 | 0
  Edema at 14 days after completion: None | 47 | 44
  Edema at 14 days after completion: Mild | 0 | 0
  Edema at 14 days after completion: Moderate | 0 | 0
  Edema at 14 days after completion: Severe | 0 | 0

4. Secondary Outcome: Change From Baseline in Sum of Participant Self-assessment Scores for Redness, Pain, Stinging/Burning, Itching, Tightness and Dryness
Description: The assessments of Pain, Stinging/ Burning, Itching, Tightness, Redness and Dryness were conducted by participants reflective of their skin condition at the 5 x 5 cm square area on the volar surface of the forearm at the time of evaluation. Participants were scored as per signs/symptom: pain, stinging/burning, itching, tightness, redness and dryness on scale of 0 to 3, where 0= none; no sign or symptoms, 1= mild; barely perceptible, 2= moderate; definite signs and symptoms, and 3= severe- marked or pronounced signs or symptoms. This outcome measure is the sum of participant scores, so a total score, i.e. the range is 0-15, with higher scores indicating increased signs or symptoms of irritation.
Time Frame: 14 days after completion of the facial peel procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 50 | 46
Score on Scale
  At Baseline | 0.38 (0.635) | 0.41 (0.805)
  14 days after completion: number analyzed (Participants) | 47 | 44
  14 days after completion | 0.02 (0.146) | 0.05 (0.211)
  Change from Baseline at 14 day after completion: number analyzed (Participants) | 47 | 44
  Change from Baseline at 14 day after completion | -0.38 (0.677) | -0.39 (0.841)

5. Secondary Outcome: Change From Baseline in Participant Self-assessment Scores for Redness
Description: The following assessments were conducted by participants reflective of their skin condition at the time of evaluation for redness. Participants were score on a scale of 0 to 3. (0= None, 1= Mild, 2= Moderate, and 3= Severe). Lower scores indicate better results.
Time Frame: 14 days after completion of the facial peel procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 50 | 46
Score on Scale
  At Baseline | 0.22 (0.507) | 0.15 (0.420)
  14 days after completion: number analyzed (Participants) | 47 | 44
  14 days after completion | 0.0 (0.00) | 0.0 (0.00)
  Change from Baseline at 14 days after completion: number analyzed (Participants) | 47 | 44
  Change from Baseline at 14 days after completion | -0.23 (0.520) | -0.16 (0.428)

6. Secondary Outcome: Change From Baseline in Participant Self-assessment Scores for Pain
Description: The following assessments were conducted by participants reflective of their skin condition at the time of evaluation for pain. Participants were scored on a scale of 0 to 3. (0= None, 1= Mild, 2= Moderate, and 3= Severe). Lower scores indicate better results.
Time Frame: 14 days after completion of the facial peel procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 50 | 46
Score on Scale
  At Baseline | 0.0 (0.00) | 0.0 (0.00)
  14 days after completion: number analyzed (Participants) | 47 | 44
  14 days after completion | 0.0 (0.00) | 00 (0.00)
  Change from Baseline at 14 days after completion: number analyzed (Participants) | 47 | 44
  Change from Baseline at 14 days after completion | 0.0 (0.00) | 0.0 (0.00)

7. Secondary Outcome: Change From Baseline in Participant Self-assessment Scores for Itching
Description: The following assessments were conducted by participants reflective of their skin condition at the time of evaluation for itching. Participants were scored on a scale of 0 to 3. (0= None, 1= Mild, 2= Moderate, and 3= Severe). Lower scores indicate better results.
Time Frame: 14 days after completion of the facial peel procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 50 | 46
Score on Scale
  At Baseline | 0.04 (0.198) | 0.02 (0.147)
  14 days after completion: number analyzed (Participants) | 47 | 44
  14 days after completion | 0.0 (0.00) | 0.02 (0.151)
  Change from Baseline at 14 days after completion: number analyzed (Participants) | 47 | 44
  Change from Baseline at 14 days after completion | -0.04 (0.204) | 0.0 (0.216)

8. Secondary Outcome: Change From Baseline in Participant Self-assessment Scores for Stinging/Burning
Description: The following assessments were conducted by participants reflective of their skin condition at the time of evaluation for stinging/burning. Participants were scored on a scale of 0 to 3. (0= None, 1= Mild, 2= Moderate, and 3= Severe). Lower scores indicate better results.
Time Frame: 14 days after completion of the facial peel procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 50 | 46
Score on Scale
  At Baseline | 0.10 (0.303) | 0.20 (0.453)
  14 days after completion: number analyzed (Participants) | 47 | 44
  14 days after completion | 0.0 (0.00) | 0.0 (0.00)
  Change from Baseline at 14 days after completion: number analyzed (Participants) | 47 | 44
  Change from Baseline at 14 days after completion | -0.11 (0.312) | -0.20 (0.462)

9. Secondary Outcome: Change From Baseline in Participant Self-assessment Scores for Tightness
Description: The following assessments were conducted by participants reflective of their skin condition at the time of evaluation for tightness. Participants were scored on a scale of 0 to 3. (0= None, 1= Mild, 2= Moderate, and 3= Severe). Lower scores indicate better results.
Time Frame: 14 days after completion of the facial peel procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 50 | 46
Score on Scale
  At Baseline | 0.0 (0.00) | 0.0 (0.00)
  14 days after completion: number analyzed (Participants) | 47 | 44
  14 days after completion | 0.0 (0.00) | 0.0 (0.00)
  Change from Baseline at 14 days after completion: number analyzed (Participants) | 47 | 44
  Change from Baseline at 14 days after completion | 0.0 (0.00) | 0.0 (0.00)

10. Secondary Outcome: Change From Baseline in Participant Self-assessment Scores for Dryness
Description: The following assessments were conducted by participants reflective of their skin condition at the time of evaluation for dryness. Participants were scored on a scale of 0 to 3. (0= None, 1= Mild, 2= Moderate, and 3= Severe). Lower scores indicate better results.
Time Frame: 14 days after completion of the facial peel procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 50 | 46
Score on Scale
  At Baseline | 0.02 (0.141) | 0.04 (0.206)
  14 days after completion: number analyzed (Participants) | 47 | 44
  14 days after completion | 0.02 (0.146) | 0.02 (0.151)
  Change from Baseline at 14 days after completion: number analyzed (Participants) | 47 | 44
  Change from Baseline at 14 days after completion | 0.0 (0.209) | -0.02 (0.263)

11. Secondary Outcome: Change From Baseline in Instrumental Measurement of Barrier Function Using Tewameter
Description: Trans-epidermal water loss (TEWL) measurement was performed by evaporimetry with a Tewameter. Measurements were taken in triplicates on the left cheek (below the cheekbone between the nose and ear). TEWL measurements were taken with the participant lying horizontally, on their back, so that the chimney of the Tewameter probe is aligned vertically. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: 14 days after completion of the facial peel procedure
Population: Analysis of TEWL was performed on Intent-to-Treat (ITT) population(N=96). Population was based on treatment to which participant was randomized. Of which, there were 50 in test product and 46 in no treatment. Here, number of participants (n=91) analyzed signifies those who were evaluated.
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 50 | 46
g/m^2/hr
  At Baseline | 20.22 (6.181) | 18.16 (4.832)
  14 days after completion: number analyzed (Participants) | 47 | 44
  14 days after completion | 17.06 (3.937) | 16.29 (3.444)
  Change from Baseline at 14 days after completion: number analyzed (Participants) | 47 | 44
  Change from Baseline at 14 days after completion | -3.37 (4.181) | -1.52 (3.571)

12. Secondary Outcome: Change From Baseline in Instrumental Measurement of Moisturisation Using Corneometer
Description: Measurement of stratum corneum hydration was performed by the electrical capacitance method with a Corneometer. Corneometer measurements were taken in triplicates at the left cheek (below the cheekbone, between the nose and ear) with the participant lying horizontally, on their back. An increase in corneometry values indicates an increase in the hydration status of the skin and vice versa.
Time Frame: 14 days after completion of the facial peel procedure
Population: Analysis of Corneometry was measured on Intent to Treat (ITT) population (N=96). Population was based on treatment to which participant was randomized. Of which, there were 50 in test product and 46 in no treatment. Here, number of participants (n=91) analyzed signifies those who were evaluated.
Measure: Mean (Standard Deviation); unit: Corneometer Units
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 50 | 46
Corneometer Units
  At Baseline | 71.39 (8.919) | 75.31 (9.718)
  14 days after completion: number analyzed (Participants) | 47 | 44
  14 days after completion | 67.09 (7.535) | 65.47 (9.279)
  Change from Baseline at 14 days after completion: number analyzed (Participants) | 47 | 44
  Change from Baseline at 14 days after completion | -4.03 (7.298) | -10.33 (10.094)

13. Secondary Outcome: Global Self-assessment of Participants
Description: Participants has rated the level of satisfaction with the post-procedure skin care regimen to which they were randomized on a scale of 0 to 3 as follows: 0 (Very satisfied), 1 (Satisfied), 2 (Poorly satisfied), 3 (Not at all satisfied). Lower scores indicate better results.
Time Frame: 14 days after completion of the facial peel procedure
Population: Global self-assessment of satisfaction was measured on ITT population (N=91). Population was based on treatment to which participant was randomized. Of which, there were 50 in test product and 46 in no treatment. Here, number of participants (n=91) analyzed signifies those who were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | No Treatment
Number analyzed (Participants) | 47 | 44
Participants
  Very Satisfied | 21 | 17
  Satisfied | 26 | 27
  Poorly Satisfied | 0 | 0
  Not at all Satisfied | 0 | 0

ADVERSE EVENTS:
Time Frame: 19 days
Description: Adverse event reporting was performed on the safety population (N=96). The safety population included all participants with at least 1 application of product in test phase. This population was based on treatment the participant actually received.
Groups:
- Test Product: Participants will apply a pea-sized quantity of test product (approximately 0.6-1 grams (g)) topically onto the fingertips and will apply twice daily (morning and evening) to the full face after cleansing. All participants will be instructed to continue using the facial cleanser twice-daily during the morning and evening and to apply the sunscreen in the morning (after application of test product) and at lunchtime.
- No Treatment: Participants will wet face with water and work a small amount of facial cleanser (approximately 0.6-1 g) into lather. Massage topically onto wet skin and rinse with water twice daily (morning and evening). After cleansing, participants will apply a pea-sized quantity (approximately 0.6-1 g) of the sunscreen in the morning and at lunchtime.
Arm/Group | Test Product | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/46
Other Adverse Events (participants affected / at risk) | 5/50 | 0/46
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=50) | No Treatment (N=46)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip Dry (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT03197883/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT03197883/SAP_001.pdf